CLINICAL TRIAL: NCT04990986
Title: Co-Development and Evaluation of a Complex Intervention to Increase Medication Safety in Nursing Homes - A Mixed Methods Study Embedding a Cluster Randomised Controlled Trial, Guided by Safety Theory With Participatory Approach
Brief Title: Co-Development and Evaluation of a Complex Intervention to Increase Medication Safety in Nursing Homes
Acronym: SAME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anne Estrup Olesen (Other)
Collaborators: Aalborg University (Other); Aalborg Municipality (Other); University College of Northern Denmark (Other)
Responsible Party: Sponsor-Investigator, Anne Estrup Olesen, Professor, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AalborgH2021-015
Record Dates: First submitted 2021-06-30; First posted 2021-08-05 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Medication Safety; Patient Safety

STUDY DESIGN:
Intervention Model Description: This study applies mixed-methods pragmatic paradigm led by Safety 1 and 2 theory, with participatory approach to an exploratory sequential three-phased study-design, embedding a randomized controlled trial (cRCT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): The complex intervention will be co-developed during first phase of the study.
  Interventions: Other: Complex intervention
- Control (No Intervention): Half of the group will be included as control and thus not exposed to the intervention.

INTERVENTIONS:
Other: Complex intervention — Will be co-developed during the study.
  Arms: Intervention

SUMMARY:
The study aims to develop and evaluate a new, multifaceted (complex) intervention in a mixed methods study-design to increase medication safety in nursing homes. The SAME-study will be locally anchored, including investigation of patient safety culture, in a mixed methods design, including both in depth qualitative and organizational-focused quantitative methods.

DETAILED DESCRIPTION:
In the SAME-study, we aim to develop and evaluate a new, multifaceted (complex) intervention in a mixed methods study-design to increase medication safety in nursing homes. The SAME-study will be locally anchored, including investigation of patient safety culture, in a mixed methods design, including both in depth qualitative and organizational-focused quantitative methods. This study will be guided by the following main research questions and hypothesis:

1. Can we elucidate new areas susceptible for intervention to increase medication safety in nursing homes through qualitative in-depth investigation of patient safety culture in nursing homes guided by safety theory with participatory approach?
2. Is it possible to develop a multifaceted intervention fit to context within actual resource-frame to increase medication safety in nursing homes based on patient safety culture, guided by safety theory with participatory approach?
3. A complex intervention developed within a participatory framework will lead to positive change of care-staff self-reported perceptions of patient safety climate culture in nursing homes in the intervention group compared with the control group of this study?

Study design This study applies mixed-methods pragmatic paradigm led by Safety 1 and 2 theory, with participatory approach to an exploratory sequential three-phased study-design, embedding a randomized controlled trial (cRCT). Overall study-settings will be nursing homes within the municipality of Aalborg, North Denmark Region, Denmark.

ELIGIBILITY:
Inclusion Criteria:

* involved directly or indirectly in the medication process
* employment of at least two months in a nursing-home within the municipality of Aalborg, sufficient spoken and written Danish language

Exclusion Criteria:

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Care staff's perceptions of patient safety culture | One year
  Safety Attitudes Questionnaire (SAQ)

SECONDARY OUTCOMES:
Perceptions of patient safety culture of relatives of residents and nursing home doctors. | One year
  Qualitative data will be collected through individual interviews with relatives and GPs

OTHER OUTCOMES:
Safety assessments | One year
  data from medical records and national registers will be used for safety assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Anne E Olesen, Ph.D., Study Director — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
We plan to publish the protocol
Supporting Information: Study Protocol
Time Frame: We plan to publish the protocol during fall 2021

REFERENCES:
- [Derived] Juhl MH, Soerensen AL, Kristensen JK, Johnsen SP, Olesen AE. Safe Medication in Nursing Home Residents Through the Development and Evaluation of an Intervention (SAME): Protocol for a Fully Integrated Mixed Methods Study With a Cocreative Approach. JMIR Res Protoc. 2023 Mar 31;12:e43538. doi: 10.2196/43538. PMID 37000508